CLINICAL TRIAL: NCT06368700
Title: The Hyalex EFS: a Prospective, Multicenter, Single-Arm, 2-Phase Early Feasibility Study (EFS) of the HYALEX® Knee Cartilage System
Brief Title: The Hyalex Early Feasibility Study (EFS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hyalex Orthopaedics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CL-00001
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Cartilage Injury; Cartilage Damage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Hyalex Knee Cartilage System (Experimental): Implantation of the Hyalex Knee Cartilage Implant
  Interventions: Device: Hyalex Knee Cartilage System

INTERVENTIONS:
Device: Hyalex Knee Cartilage System — Surgical implantation of the Hyalex Knee Cartilage System

SUMMARY:
The Hyalex Early Feasibility Study is a prospective, multicenter, open-label, single-arm, 2-phase early feasibility study to evaluate the safety and technical performance of the HYALEX Knee Cartilage System for replacement of loss of articular cartilage and bone of the knee femoral condyles in symptomatic patients who require surgical treatment, will be enrolled in the study and undergo implantation of the HYALEX Knee Implant.

ELIGIBILITY:
Inclusion Criteria (Phase 1):

1. 21-70 years.
2. Body Mass Index (BMI) ≤ 38.
3. Singular treatable joint surface lesion, ICRS Grade 3 or 4, located on the medial or lateral femoral condyle.
4. One implant to treat a single symptomatic lesion with up to 3.8cm2 total lesion area.
5. Knee Injury and Osteoarthritis Outcome Score (KOOS) pain subscale score between 20 and 65.
6. Stable knee.
7. Failure of non-operative treatment (e.g., physical therapy, physician-directed at home exercise program, intra-articular injections, bracing) for at least 4 weeks prior to consideration for participation in the study.

Inclusion Criteria (Phase 2):

1. 21-70 years.
2. Body Mass Index (BMI) ≤ 38.
3. Up to three treatable joint surface lesion(s), ICRS Grade 3 or 4, located on the medial or lateral femoral condyle(s).
4. Up to 3 implants to treat up to 3 individual symptomatic lesions with a total summative area up to 10cm2.
5. Knee Injury and Osteoarthritis Outcome Score (KOOS) pain subscale score between 20 and 65.
6. Stable knee.
7. Failure of non-operative treatment (e.g., physical therapy, physician-directed at home exercise program, intra-articular injections, bracing) for at least 4 weeks prior to consideration for participation in the study.

Exclusion Criteria:

HYALEX Implant, Surgical Technique, and Lesion Site Exclusions:

1. Known allergy to polyurethanes, bone cement, acrylic, or titanium.
2. Lack of 2mm of healthy cartilage (ICRS Grade 0 to 2) and 2mm of vital bone wall on all sides of the implant site.
3. Osteochondral defect affecting subchondral bone more than 11mm in depth from adjacent non-defect articular surface.
4. Bipolar cartilage lesions involving patellar or tibial lesions ICRS Grade 3 - 4 opposite the lesion intended for treatment.
5. Insufficient bone stock or bone density determined intra-operatively preventing implant press fit.

Patient Orthopaedic Health Exclusions:

1. Kellgren and Lawrence (KL) grade 3 or 4 on standing radiographs.
2. Hip-knee-ankle (HKA) angle of greater than +/- 8 degrees (varus or valgus malalignment > 8 degrees) on standing X-ray.
3. Lack of normally functioning contralateral knee that restricts activity.
4. Insufficiency fracture of the femoral condyle or tibial plateau.
5. Recent Osteochondritis Dissecans within 1 year.
6. Diagnosis of a concomitant knee injury which the investigator believes may interfere with study participation or confound effectiveness assessment.
7. Untreated ACL and/or PCL deficiency or complex ligamentous instability of the study knee according to IKDC Grade C (abnormal) or D (severely abnormal).

Previous Surgery and Intervention Exclusions:

1. Previous surgical cartilage treatment in the index knee within the last 6 months
2. Previous intra-articular injections, including HA and steroids, within the last 3 months prior to the date of surgery.

Patient Overall Health and Health History Exclusions:

1. Any known history of inflammatory arthropathy or crystal-deposition arthropathy.
2. Current cigarette smoker or user of other nicotine products.
3. Known Type 1 or Type 2 insulin-dependent diabetes mellitus.
4. Currently undergoing immunosuppressive therapy or long-term steroid use (corticosteroid, excluding inhalers) or within 3 months prior to surgery.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Freedom from implant rejection and infection. | 12 months
  To assess the safety (implant rejection, implant dislocation or disassociation (delamination), infection) and tolerability of the Hyalex Knee Cartilage Implant.
Change in the Knee Injury & Osteoarthritis Outcome Score (KOOS) at 12 months. | 12 months
  The KOOS assesses patient pain, other symptoms, function in daily living, function in sport and recreation, and knee related quality of life. Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Horizon Clinical Research, La Mesa, California
  - Ochsner Sports Medicine Institute, New Orleans, Louisiana
  - Hospital for Special Surgery, New York, New York
  - Oregon Health & Science University, Portland, Oregon